CLINICAL TRIAL: NCT00217646
Title: Phase I Study of BAY 43-9006 (NSC 724772) in Patients With Acute Leukemias, Myelodysplastic Syndromes and Chronic Myeloid Leukemia in Blast Phase
Brief Title: Sorafenib in Treating Patients With Refractory or Relapsed Acute Leukemia, Myelodysplastic Syndromes, or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00081; NCI-2009-00081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000442847; 2004-0702 (Other: M D Anderson Cancer Center); 6742 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2013-02

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Acute Promyelocytic Leukemia With t(15;17)(q22;q12); PML-RARA; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Blastic Phase; de Novo Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Sorafenib

ARMS (2):
- Arm I (Experimental): Patients receive oral sorafenib once or twice daily on days 1-5, 8-12, and 15-19.
  Interventions: Drug: Sorafenib Tosylate
- Arm II (Experimental): Patients receive oral sorafenib once or twice daily on days 1-14.
  Interventions: Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of two different schedules of sorafenib in treating patients with refractory or relapsed acute leukemia, myelodysplastic syndromes, or blastic phase chronic myelogenous leukemia. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of sorafenib when administered in two different schedules in patients with refractory or relapsed acute leukemia, myelodysplastic syndromes, or blastic phase chronic myelogenous leukemia.

II. Determine the dose-limiting toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this drug in these patients. II. Determine the biologic effect of this drug in these patients.

OUTLINE: This is a randomized, dose-escalation phase I study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral sorafenib once or twice daily on days 1-5, 8-12, and 15-19.

Arm II: Patients receive oral sorafenib once or twice daily on days 1-14.

In both arms, treatment repeats every 21 days for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission or partial remission after 6 months may continue therapy at the discretion of the principal investigator.

In both arms, cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 patients are treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following: Acute myeloid leukemia (Acute promyelocytic leukemia (M3) allowed provided patient has failed prior therapy with both tretinoin and arsenic alone or in combination); Acute lymphoblastic leukemia; Myelodysplastic syndromes; Blastic phase chronic myelogenous leukemia (Failed OR intolerant to imatinib mesylate)
* Must have failed prior therapy with >= 1 cytotoxic- or biologic-targeted agent (e.g., hypomethylating agents, farnesyl transferase inhibitors, thalidomide, or tyrosine kinase inhibitors); Any number of prior regimens allowed
* Performance status: ECOG 0-1
* ALT =< 2.5 times upper limit of normal
* Bilirubin =< 1.5 mg/dL
* Creatinine =< 2.0 mg/dL OR Creatinine clearance >= 60 mL/min
* Fertile patients must use effective contraception
* No psychiatric illness or social situation that would preclude study compliance
* Prior bone marrow transplantation allowed
* At least 2 weeks since prior cytotoxic agents OR at least 5 half-lives for non-cytotoxic agents in the absence of rapidly progressing disease
* At least 24 hours since prior hydrea for control of peripheral blood leukemia cell counts
* Hydroxyurea allowed up to 72 hours after start of therapy with sorafenib
* No persistent, chronic, clinically significant toxicities > grade 1 from prior chemotherapy

Exclusion Criteria:

* Cytopenias secondary to multilineage bone marrow failure allowed
* Ineligible for or not willing to undergo allogeneic stem cell transplantation OR no donor available
* Absolute blast count=< 20,000/mm^3 unless patient has documented fms-like tyrosine kinase 3 internal tandem duplication
* No evidence of bleeding diathesis (except due to low platelets associated with the primary disease)
* No New York Heart Association class III or IV congestive heart failure
* No uncontrolled hypertension (i.e., sustained systolic blood pressure [BP] >= 150 mm Hg or diastolic BP >= 90 mm Hg)
* No unstable angina pectoris
* No symptomatic cardiac arrhythmia requiring and not responding to medical intervention
* Not pregnant or nursing
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to the study drug
* No swallowing dysfunction that would impede oral ingestion of tablets
* No active uncontrolled infection
* No other uncontrolled illness
* No prior sorafenib
* No other concurrent investigational or commercial agents, except for standard intrathecal chemotherapy for the treatment of isolated CNS leukemic involvement
* No other concurrent anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic anticoagulation (Concurrent prophylactic anticoagulation [i.e., low-dose warfarin, catheter flushing with heparin] of venous or arterial access devices allowed)
* No concurrent cytochrome P450 enzyme-inducing antiepileptic agents, including, but not limited to, any of the following: Phenytoin; Carbamazepine; Phenobarbital; Rifampin
* No concurrent Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Borthakur G, Kantarjian H, Ravandi F, Zhang W, Konopleva M, Wright JJ, Faderl S, Verstovsek S, Mathews S, Andreeff M, Cortes JE. Phase I study of sorafenib in patients with refractory or relapsed acute leukemias. Haematologica. 2011 Jan;96(1):62-8. doi: 10.3324/haematol.2010.030452. Epub 2010 Oct 15. PMID 20952518